CLINICAL TRIAL: NCT06963281
Title: A Phase 1, Multicenter, Open-label Study of IBI3020 Treatment in Participants With Unresectable, Locally Advanced or Metastatic Solid Tumors
Brief Title: Study of IBI3020 Treatment in Participants With Late-Stage Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biopharmaceutical Technology (Hangzhou) Co., LTD. (Industry)
Collaborators: Fortvita Biologics (USA)Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: "CIBI3020A101"
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- IBI3020 (Experimental)
  Interventions: Drug: IBI3020

INTERVENTIONS:
Drug: IBI3020 — Recombinant anti-CEACAM5 monoclonal antibody - dual-payload conjugate for injection

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of IBI3020 and to determine the maximum tolerated dose (MTD) and/or the recommended dose for expansion (RP2D) of IBI3020.

ELIGIBILITY:
Inclusion Criteria:

Participants must satisfy all of the following criteria to be enrolled into the study:

1. Participants have the ability to understand and give written informed consent for participation in this trial, including all evaluations and procedures as specified by this protocol;
2. Male or female participants ≥ 18 years old. For Part 1, age ≥ 18 years and ≤ 75 years;
3. Histologically or cytologically confirmed unresectable, locally advanced or metastatic solid tumors which have received available standard therapies and have disease progression, or unacceptable toxic effects, or contraindications;
4. At least 1 measurable lesion as defined per RECIST v1.1 within 28 days prior to the first dose of IBI3020;
5. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0-1;
6. Minimum life expectancy of 12 weeks;
7. Adequate bone marrow and organ function confirmed at screening period;
8. Participants, both male and female, who are not of childbearing potential or who agree to use at least 1 highly effective method of contraception during the study.

Exclusion Criteria:

Participants who meet any of the following criteria will be disqualified from entering the study:

1. Previous treatment with CEACAM5-targeted therapy;
2. Prior anti-cancer therapy within the wash-out period;
3. Received live vaccines within 4 weeks or cancer vaccine within 3 months;
4. Potent cytochrome P450 3A4 (CYP3A4) inhibitors within 2 weeks or 5 half-lives;
5. Has adverse reactions resulting from previous anti-tumor therapies, which have not resolved to Grade 0 or 1 toxicity according to NCI CTCAE v5.0;
6. Known allergies, hypersensitivity, or intolerance to IBI3020 or its excipients;
7. Undergone major surgery within 4 weeks, or who have severe unhealed wounds;
8. Known symptomatic central nervous system (CNS) metastases;
9. Uncontrolled diseases or conditions;
10. History of pneumonitis requiring corticosteroids therapy, or history of clinically significant lung diseases;
11. History of thromboembolic event within 6 months;
12. Under neurological, psychiatric or social condition;
13. Women who are pregnant, have positive results in pregnancy test or are lactating;
14. Not eligible to participate in this study at the discretion of the investigator;
15. Participating in any other interventional clinical research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Numbers of subjects with adverse events | Up to 3 years
  defined as any untoward medical occurrence, whether or not there is a causal relationship with the study drug, in a clinical study subject from the time informed consent form is signed
Number of subjects with clinically significant changes in physical examination results | Up to 3 years
  Clinically significant abnormal physical examination findings reported by the investigator.
Number of subjects with clinically significant changes in electrocardiogram | Up to 3 years
  Clinically significant abnormal electrocardiogram findings reported by the investigator.
Number of subjects with clinically significant changes in vital signs | Up to 3 years
  Vital signs including body temperature, pulse, respiratory rate, oxygen saturation by pulse oximetry at rest and blood pressure
Dose limiting toxicities (DLTs) | Up to 21 days
  Dose limiting toxicities (DLTs) to establish MTD and/or RP2D.
objective response rate (ORR) | Up to 3 years
  objective response rate (ORR) as evaluated per the RECIST v1.1 criteria.
Number of subjects with clinically significant changes in laboratory parameters | Up to 3 years
  Clinically significant abnormal laboratory parameters findings reported by the investigator.

SECONDARY OUTCOMES:
area under the curve (AUC) | Up to 3 years
  area under the curve (AUC) of single and multiple doses of IBI3020
maximum concentration (Cmax) | Up to 3 years
  maximum concentration (Cmax) of single and multiple doses of IBI3020
time to maximum concentration (Tmax) | Up to 3 years
  time to maximum concentration (Tmax) of single and multiple doses of IBI3020
clearance (CL) | Up to 3 years
  clearance (CL) of single and multiple doses of IBI3020
apparent volume of distribution (V) | Up to 3 years
  apparent volume of distribution (V) of single and multiple doses of IBI3020
half-life (t1/2) | Up to 3 years
  half-life (t1/2) of IBI3020 to the last administration of IBI3020
anti-drug antibody (ADA) | Up to 3 years
  Incidence and characterization of anti-drug antibody (ADA).
objective response rate (ORR) | Up to 3 years
  objective response rate (ORR) as evaluated per the RECIST v1.1 criteria.
duration of response (DoR) | Up to 3 years
  duration of response (DoR) as evaluated per the RECIST v1.1 criteria.
time to response (TTR) | Up to 3 years
  time to response (TTR) as evaluated per the RECIST v1.1 criteria.
progression free survival (PFS) | Up to 3 years
  as evaluated per the RECIST v1.1 criteria.
disease control rate (DCR) | Up to 3 years
  disease control rate (DCR)as evaluated per the RECIST v1.1 criteria.
overall survival (OS) | From date of randomization until the date of first documented date of death from any cause, assessed up to 36 months
  OS is defined as the time from the date of first dose of study drug until the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (6):
  - Mayo Clinic - Arizona, Pheonix, Arizona
  - Mayo Clinic - Florida, Jacksonville, Florida
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Montefiore Cancer Center, New York, New York
  - NEXT Houston, Houston, Texas
  - NEXT Dallas, Irving, Texas
- China (3):
  - The sixth affiliated hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanxi Cancer Hospital, Taiyuan, Shanxi